CLINICAL TRIAL: NCT07342673
Title: Vital Coach: A Study of Resiliency in Medical Students Using Wearable Technology and Personalized Wellness Coaching
Brief Title: Vital Coach: A Study of Resiliency in Medical Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00140462
Record Dates: First submitted 2025-12-08; First posted 2026-01-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Burnout
Keywords: wellness coaching; performance coaching; biometric feedback; psychological stress
MeSH Terms: conditions — Burnout, Psychological; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: first-year medical students from Wake Forest School of Medicine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arena Strive (Experimental): digital coaching platform, which integrates asynchronous coaching, two virtual coaching sessions with a high-performance medicine coach, physiological data from wearable sensors, and a focused curriculum of performance tools tailored to frontline healthcare workers.
  Interventions: Behavioral: Arena Strive

INTERVENTIONS:
Behavioral: Arena Strive — integrates asynchronous coaching, two virtual coaching sessions with a high-performance medicine coach, physiological data from wearable sensors, and a focused curriculum of performance tools tailored to frontline healthcare workers.
  Other Names: digital coaching platform

SUMMARY:
Medical students often begin training with psychological and physiological health metrics superior to their age-matched peers. By graduation, however, rates of depression, anxiety, and physiologic dysregulation are markedly higher, reflecting the cumulative strain of long study hours, high-stakes examinations, and the emotional burden of early patient care. Despite this, few medical schools provide structured, evidence-based tools for students to develop resiliency and recovery skills before clinical rotations begin.

DETAILED DESCRIPTION:
This gap represents both a health crisis and an educational opportunity. Burnout originating in medical school often persists into residency and practice, diminishing empathy and professionalism, and contributing to long-term attrition. Existing wellness offerings are largely reactive, relying on voluntary counseling or broad wellness sessions that fail to provide individualized insight into students' physiological readiness or stress recovery capacity. Moreover, schools lack objective, continuous data to pinpoint when students are physiologically stressed to tailor timely support.

Against this backdrop, this study proposes evaluating a structured performance coaching and biometric feedback approach in the context of scheduled academic stressors. Arena Strive is a digital coaching platform that integrates a virtual human performance coach, wearable-derived biometric data, and a focused skills curriculum adapted from other high-stress domains and tailored to frontline healthcare workers. This novel intervention has proven effective in significantly reducing burnout and enhancing professional fulfillment and self-valuation in a large health-system through an 8-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* active first year Wake Forest School of Medicine medical students
* have an Android or iOS smart phone
* are willing to download the Arena Strive application

Exclusion Criteria:

* under the age of 18; or over the age of 60
* pregnant at enrollment or during course of study
* any self-reported cardiac conditions that may impact heart rate and heart rate variability

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability | Weekly through Week 13
  Mean daily nocturnal Heart Rate Variability (HRV): Higher = Better
Resting Heart Rate (Beats per Minute) | Weekly through Week 13
  daily nocturnal Resting Heart Rate (RHR): Lower = Better
Sleep Duration (minutes) | Weekly through Week 13
  Mean nightly sleep: Higher = Better
Sleep Consistency (minutes) | Weekly through Week 13
  SD of mid-sleep time: Lower = Better

SECONDARY OUTCOMES:
Change in Perceived Stress (Perceived Stress Scale PSS-4) Scores | Weekly through Week 13
  To score the Perceived Stress Scale 4 (PSS-4), first, reverse the scores for questions 2 and 3 (0 becomes 4, 1 becomes 3, 2 stays 2, 3 becomes 1, and 4 becomes 0). Then, add up the scores for all four questions. The total score will range from 0 to 16, with higher scores indicating greater perceived stress.
Change in Burnout (Maslach Burnout Inventory MBI-GSS) Scores | Week 13
  MBI-GSS scoring involves summing responses for each of its three subscales: emotional exhaustion, cynicism, and professional efficacy, which are rated on a 7-point frequency scale from 0 (never) to 6 (daily). To determine burnout, high scores on exhaustion and cynicism indicate higher burnout, while low scores on professional efficacy suggest greater burnout. These subscale scores are then interpreted separately to understand the level of burnout for each dimension. Each item is rated on a frequency scale (e.g., 0 to 6), and higher or lower scores on each subscale indicate different levels of burnout.

OTHER OUTCOMES:
Exam Performance checklist | Week 13
  Exam performance for the three exams during the study period is self-reported by participants via a typeform in the application at the study conclusion.
Weekly mean nocturnal HRV (RMSSD, ms) measured via wearable device during intervention and compared to other phases. | Weekly through Week 13
  HRV will be assessed using the root mean square of successive differences (RMSSD, ms) to provide a daily individual score derived from nightly photoplethysmography (PPG) wearable-recorded data. All primary endpoints are computed at the individual level and compared by week, using week-level means (averaged from the individual daily scores). Heart Rate Variability (HRV) [RMSSD, ms] Individual Test= Like earlier mentioned tests these will include week-to-week differences for the weeks during the phase (Baseline Week, Study Week, Exam Week, Recovery Week) (ex. HRV_Recovery (during) - HRV_Exam (during) and comparisons with pre/post intervention phases (ex. HRV_Recovery (during) - HRV_Recovery (pre-intervention)).
  Group Test= A linear mixed model for HRV and PSS-4 with fixed effects for Week, Phase (0=pre, 1=post, 2=during) and a Week x Phase interaction, plus a random intercept for participant.
  Sensitivity Analyses= Paired t-tests (Wilcoxon as nonparametric alternative).
Weekly mean nocturnal RHR (bpm) measured via wearable device during intervention and compared to other phases. | Weekly through Week 13
  Daily mean RHR (bpm) will be derived from nightly PPG wearable-recorded data. All primary endpoints are computed at the individual level and compared by week using week-level means (averaged from the individual daily scores). Resting Heart Rate (RHR) [bpm] Individual Test= Like earlier mentioned tests these will include week-to-week differences for the weeks during the phase (Baseline Week, Study Week, Exam Week, Recovery Week) (ex. RHR_Recovery (during) - RHR_Exam (during) and comparisons with pre/post intervention phases (ex. RHR_Recovery (during) - RHR_Recovery (pre-intervention)).
  Group Test= A linear mixed model for RHR and PSS-4 with fixed effects for Week, Phase (0=pre, 1=post, 2=during) and a Week x Phase interaction, plus a random intercept for participant.
  Sensitivity Analyses= Paired t-tests (Wilcoxon as nonparametric alternative).
Weekly mean Sleep Duration (min) measured via wearable device during intervention and compared to other phases. | Weekly through Week 13
  Daily Sleep Duration (min) will be derived from nightly PPG wearable-recorded data. All primary endpoints are computed at the individual level and compared by week using week-level means (averaged from the individual daily scores). Sleep Duration [min] Individual Test= Like earlier mentioned tests these will include week-to-week differences for the weeks during the phase (Baseline Week, Study Week, Exam Week, Recovery Week) (ex. SleepDuration_Recovery (during) - Sleep Duration_Exam (during) and comparisons with pre/post intervention phases (ex. SleepDuration_Recovery (during) - SleepDuration_Recovery (pre-intervention)).
  Group Test= A linear mixed model for Sleep Duration and PSS-4 with fixed effects for Week, Phase (0=pre, 1=post, 2=during) and a Week x Phase interaction, plus a random intercept for participant.
  Sensitivity Analyses= Paired t-tests (Wilcoxon as nonparametric alternative).
Weekly Sleep Consistency (SD of mid-sleep time, min) measured via wearable device during intervention and compared to other phases. | Weekly through Week 13
  Sleep Consistency will be measured as the standard deviation of nightly mid-sleep time derived from wearable-recorded sleep onset and offset times over each 7-day period, aggregated weekly at the individual level and compared across pre-intervention, intervention, and post-intervention phases. Sleep Consistency Individual Test= Like earlier mentioned tests these will include week-to-week differences for the weeks during the phase (Baseline Week, Study Week, Exam Week, Recovery Week) (ex. SleepConsistency_Recovery (during) - SleepConsistency_Exam (during) and comparisons with pre/post intervention phases (ex. SleepConsistency_Recovery (during) - SleepConsitency_Recovery (pre-intervention)).
  Group Test= A linear mixed model for Sleep Consistency and PSS-4 with fixed effects for Week, Phase (0=pre, 1=post, 2=during) and a Week x Phase interaction, plus a random intercept for participant.
  Sensitivity Analyses= Paired t-tests (Wilcoxon as nonparametric alternative).
Heterogeneity of effects (sensitivity only) | Weekly through Week 13
  Moderation by demographics (age, race, gender) on primary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Dermot Phelan, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No